CLINICAL TRIAL: NCT01403285
Title: A Phase 1 Trial of Peptide-Based Glioma Vaccine IMA950 in Patients With Glioblastoma (GBM)
Brief Title: Peptide-based Glioma Vaccine IMA950 in Patients With Glioblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to poor accrual. This decision was taken without any safety reasons. Since beginning of the study (June 2011) only six patients were enrolled.
Sponsor: Immatics Biotechnologies GmbH (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMA950-102; 11C0192 (Other: National Cancer Institute); NCT01386463 (obsolete NCT alias)
Record Dates: First submitted 2011-07-21; First posted 2011-07-27 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; stable disease
MeSH Terms: conditions — Glioblastoma | interventions — Cyclophosphamide; IMA950; Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors; sargramostim; Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cyclophosphamide — One single low-dose i.v. infusion of cyclophosphamide (300mg/m2) prior to the first vaccination as pre-treatment
  Other Names: - Cytoxan (US name); - Endoxan (EU name)
Biological: IMA950 plus GM-CSF — Six vaccinations with IMA950 plus GM-CSF as adjuvant on 8 pre-defined days from Day 1 to Day 78
  Other Names: - Granulocyte macrophage-colony stimulating factor; - Sargramostim; - Leukine
Biological: IMA950 — After Day 78, vaccinations with IMA950 (no GM-CSF) will be given on a monthly basis for up to one year from start of vaccination or until disease progression
Drug: Imiquimod — Imiquimod will be topically applied 10-20 minutes after each vaccination. After the third vaccination onward patients will apply additional imiquimod 24 hours after each vaccination at home on their own
  Other Names: - Aldara

SUMMARY:
BACKGROUND: Active immunotherapy of cancer is based on the premise that the vaccine raises a cytotoxic immune response to tumor-associated antigens, thereby destroying malignant cells without harming normal cells.

IMA950 is a therapeutic multi-peptide vaccine containing 11 tumor-associated peptides (TUMAPs) found in a majority of glioblastomas, and is designed to activate TUMAP-specific T cells. The use of 11 TUMAPs increases the likelihood of a multi-clonal, highly specific T-cell response against tumor cells leading to decreased likelihood of immune evasion of the tumor by down-regulation of target antigens.

PURPOSE: The primary objective of this study is to determine the safety and tolerability of IMA950 when given with cyclophosphamide, granulocyte macrophage-colony stimulating factor (GM-CSF) and imiquimod in patients with glioblastoma and to determine if IMA950 shows sufficient immunogenicity in these patients.

ELIGIBILITY: Patients with histologically proven GBMs who have completed radiotherapy, and have stable disease following at least 4 cycles of adjuvant temozolomide.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven glioblastoma
* Stable disease following ≥ 4 cycles of adjuvant temozolomide
* No progression or recurrence of disease

PATIENT CHARACTERISTICS:

* HLA-A*02 positive
* ≥ 18 years old
* Life expectancy > 8 weeks
* Karnofsky performance status ≥ 60
* WBC >3,500/µL
* ALC >350/mm3
* ANC >1,500/mm3
* Platelet count >100,000/mm3
* Hemoglobin >10gm/dL
* AST, ALT and alkaline phosphatase <2.5 times upper limit of normal (ULN)
* Bilirubin <1.5 times ULN
* Creatinine <1.5 mg/dL and/or creatinine clearance >60cc/min
* Serum potassium, magnesium and calcium within normals levels (supplementation is allowed)
* Not pregnant or nursing
* Negative pregnancy test
* Practice birth control during and for 2 months after treatment with IMA950 (both genders)
* Women of childbearing age must agree to use adequate contraceptive methods
* No significant active hepatic, renal, infectious or psychiatric disease
* No HIV, active hepatitis infection, or any other active severe infectious disease
* No history of autoimmune disease or immunosuppression
* No clinically significant cardiovascular event within 3 months before study entry or an increased risk for ventricular arrhythmia
* No malignancy other than glioblastoma that required treatment during the last 12 months

PRIOR and/or CONCURRENT THERAPY:

* See Disease Characteristics
* Completed radiotherapy and at least 4 cycles of adjuvant temozolomide
* Not be receiving steroids OR be on stable dose of steroids for ≥ 5 days prior to registration
* No other prior immunotherapy for glioblastoma
* No major surgery within 4 weeks prior to treatment start
* At least 4 weeks from cytotoxic therapies (incl. temozolomide)
* At least 2 weeks from non-cytotoxic therapies (e.g. interferon, tamoxifen)
* At least 3 weeks from bevacizumab
* No current treatment with imiquimod; prior use of imiquimod is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of IMA950 administered with granulocyte macrophage colony stimulating factor (GM-CSF) and topical imiquimod together following a single low-dose application of cyclophosphamide. | Continuously for up to 1 year plus follow-up
  Number of AEs and percentage of patients with AEs (listed per grade and MedDRA preferred terms) will be reported.
Immunogenicity of IMA950 | 6 time points (blood drawings) during the first 3 months (pre- and post-vaccination)
  Vaccine-induced immune responses to peptides contained in IMA950 will be measured by multimer assay using peripheral blood. Percentage of immune responders (patients with at least one vaccine-induced immune response to IMA950 peptides) and percentage of multi-TUMAP responders (patients with vaccine-induced immune responses to ≥2 peptides in IMA950) will be reported.

SECONDARY OUTCOMES:
Immune status parameters | 6 time points (blood drawings) during the first 3 months on study (pre-vaccination and during vaccination period)
  Relative frequencies and absolute numbers per µl blood of regulatory T-cells and (if sufficient cells are available) other immune cell populations will be measured from peripheral blood. Focus is on analysis of pre-vaccination frequencies.
Biomarker assessment and correlation to clinical and immunological response | Analysis time points are before the first vaccination and 15 weeks thereafter
  Serum levels of proteins and other factors that are indicative of the immune status of the patients will be measured (e.g TGF-beta) and will be correlated with immune response rates and clinical outcome.
Clinical anti-tumor activity (response rate, 6-month progression-free survival) | Will be followed for 1 year (until end of study visit), overall survival will also be followed thereafter
  Clinical response rates, survival and progression-free survival (PFS) will be followed. PFS at 6 month will be reported.
Influence of corticosteroids on immunogenicity of IMA950 | 6 time points (blood drawings) during the first 3 months (pre- and post-vaccination)
  Corticosteroid levels are not limited in this trial. It will descriptively reported whether the known immunosuppressive effects of corticosteroids are reflected in different immune response rates for patients treated or not treated with corticosteroids.
Health-related quality of life | Monthly for 1 year
  FACT-Br(4.0) questionnaire will be used to assess HRQL. HRQL scores (total, Trial Outcome Index, subscales) will be reported at baseline. Changes from baseline will also be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Teri Kreisl, MD, Principal Investigator — Neuro-Oncology Branch of the National Cancer Institute, National Institutes of Health, Bethesda, MD
Locations (1):
- Neuro-Oncology Branch of the National Cancer Institute, National Institutes of Health, Bethesda, Maryland, United States